CLINICAL TRIAL: NCT01482923
Title: Feasibility of Tobacco Assessment and Intervention With Low-Income Persons Living With HIV-AIDS (PLWHA) in Community-Based AIDS Service Organizations
Brief Title: Tobacco Assessment and Intervention With Low-Income Persons Living With HIV-AIDS (PLWHA) in Community-Based AIDS Service Organizations
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Gay Men's Health Crisis (Unknown); The City College of New York (Other); AIDS Center of Queens County (Unknown); Bronx AIDS Services (Unknown); North Jersey Community Research Initiative (Other)
Responsible Party: Sponsor
Other Study IDs: 11-173
Record Dates: First submitted 2011-11-28; First posted 2011-12-01 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Tobacco Cessation; HIV; AIDS
Keywords: Tobacco Use Assessment; smoke tobacco; quit smoking; tobacco cessation; HIV/AIDS; Community-Based Service Organizations; 11-173; Low-Income Persons Living with HIV/AIDS
MeSH Terms: conditions — Tobacco Use Cessation; Acquired Immunodeficiency Syndrome | interventions — Therapeutics; Air; Inhalation; Respiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Treatment As Usual (TAU): This study is a pilot intervention trial examining the feasibility of a motivational smoking cessation intervention using respiratory biomarker feedback in low income PLWHA. The plan is to recruit a pilot sample of 50 eligible and consented participants, randomized at a 1:1 ratio into either the Treatment As Usual (TAU) condition or the experimental (Aspiration, Inspiration Respiration, or AIR) intervention condition.
  Interventions: Behavioral: Treatment as usual
- Aspiration, Inspiration Respiration, or AIR: This study is a pilot intervention trial examining the feasibility of a motivational smoking cessation intervention using respiratory biomarker feedback in low income PLWHA. The plan is to recruit a pilot sample of 50 eligible and consented participants, randomized at a 1:1 ratio into either the Treatment As Usual (TAU) condition or the experimental (Aspiration, Inspiration Respiration, or AIR) intervention condition.
  Interventions: Behavioral: AIR (Aspirations, Inspiration, Respiration)

INTERVENTIONS:
Behavioral: Treatment as usual — Participants in the Treatment as Usual study arm will be provided with the following: 1) brief smoking cessation counseling as recommended in the Public Health Service treatment guidelines; 2) direct referral to the NY/NJ State Quitline; 3) a brochure that describes the Quitline services and provides contact information via telephone or internet; 4) a NY State brochure on HIV and smoking that identifies the specific risks of smoking for PLWHA; and 5) referral assistance to participants who present with untreated co-morbid conditions.
  Groups: Treatment As Usual (TAU)
Behavioral: AIR (Aspirations, Inspiration, Respiration) — Participants in the Aspirations, Inspiration, and Respiration study arm will receive all of the components of Treatment as Usual along with these additional components: 1) a lung age test to determine the ability and functioning of their lungs; 2) a personal lung health report with their lung age, the CO level of their breath, and a summary of their respiratory symptom assessment; 3) a review of this personal lung health report with a study counselor, 4) motivational interviewing techniques guided by Self-Determination Theory concepts to explicitly elicit at least one life aspiration of the patient and encourage discussion of such aspirations using an autonomy-supportive approach.
  Groups: Aspiration, Inspiration Respiration, or AIR

SUMMARY:
"A treatment session especially for PLWHA to help them discuss and take action about their smoking may be useful."

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older as per self-report;
* English speaking;
* New York or New Jersey State resident;
* HIV-positive serostatus direct referral from a CAB agency staff member, which verifies that the person is an HIV+ client, or by as verified by presentation of medical evidence (i.e.,confirmatory test result, ARV prescription, M11Q form, or lab results);
* Self-report of smoking > or = to 20 cigarettes (> or = to one pack) within the prior 7 days;
* To confirm smoking status, the carbon monoxide alveolar breath test must be > or = to 10 ppm;
* To confirm cognitive functioning, score on the in-person BLESSED Exam must be < or = to 10;
* Low income, defined by either: 1) Proof of Medicaid insurance, or 2) Self-report of income at 50% or below median income for New York State for New York State residents, or if a New Jersey resident, at or below 50% median income for New Jersey

Exclusion Criteria:

* Presence of current severe psychopathology that would limit study participation (e.g., unstable schizophrenia, bipolar disorder recent changes to medication noncompliance);
* Currently receiving smoking cessation treatment elsewhere.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: "Low-income smokers living with HIV/AIDS being served at community-based organizations."
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2011-11-22 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of a motivational tobacco cessation intervention | 2 years
  The study will test whether the percentage of eligible and enrolled study participants who complete the assigned intervention is significantly different from a population of percentages centered at 45%, i.e., the "null population percentage," considered a percentage too low to be compatible with feasibility."

SECONDARY OUTCOMES:
Estimate the differences between the experimental intervention | 2 years
  Assess potential factors influencing study participation by community organizations" and, as the description, "Descriptive statistics will be summarized by participating community organizations on each organization's "Implementation Factors" assessment, an agency study participation measure developed for this project. The measure assesses how many clients the agency has referred, what means were used to recruit, and what barriers to recruitment were encountered, and an open-ended question is provided for additional input."

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- City College of New York, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/